CLINICAL TRIAL: NCT07257666
Title: The Effect of Platelet-rich Fibrin on the Regeneration of Patellar Ligament Defects and the Functional Recovery of Patients After Anterior Cruciate Ligament Reconstruction of the Knee
Brief Title: Sensory Deficit Following ACL Reconstruction: PRF Pilot Study
Acronym: PRF-ACL
Status: Completed | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Darko Milovanovic, Principal Investigator, University Clinical Center of Serbia, Docent, Faculty of Medicine, University of Belgrade, University of Belgrade
Other Study IDs: Eticka komisija 17/VI-3; 17/VI-3 (Other: Ethics Committee of the Faculty of Medicine, University of Belgrade - Approval No. 17/VI-3)
Record Dates: First submitted 2025-09-23; First posted 2025-12-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Anterior Cruciate Ligament Injury; Knee Injuries; Sensory Disorders; Bone-Patellar Tendon-Bone Autograft; Platelet-Rich Fibrin (PRF)
Keywords: Platelet-Rich Fibrin; ACL reconstruction; Bone-Patellar Tendon-Bone autograft; Anterior Cruciate Ligament Injury; Knee Surgery; Sensory Deficit; Donor Site Morbidity
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries; Sensation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PRF Group: Patients undergoing ACL reconstruction with a bone-patellar tendon-bone (BPTB) autograft, with platelet-rich fibrin (PRF) applied at the donor site (n=24)
  Interventions: Biological: Platelet-rich fibrin (PRF)
- Control Group: Patients undergoing ACL reconstruction with a BPTB autograft, treated with standard closure without PRF (n=29)
  Interventions: Procedure: Standard Closure (Control)

INTERVENTIONS:
Biological: Platelet-rich fibrin (PRF) — Autologous PRF prepared intraoperatively from patient's venous blood and applied at the donor site after graft harvesting.
  Other Names: Autologous PRF
  Groups: PRF Group
Procedure: Standard Closure (Control) — Conventional closure of the donor site without PRF application
  Groups: Control Group

SUMMARY:
Pilot, single-center, non-randomized, parallel-group clinical study designed to assess whether intraoperative application of autologous platelet-rich fibrin (PRF) at the bone-patellar tendon-bone (BPTB) donor site reduces postoperative anterior knee sensory deficit after anterior cruciate ligament (ACL) reconstruction in competitively active male athletes. Planned enrollment is 53 participants allocated to a PRF cohort or a standard-care cohort. The primary outcome is the proportion of participants without anterior knee sensory deficit at 12 months post-surgery.

DETAILED DESCRIPTION:
Background: Sensory deficit around the BPTB donor site is a recognized complication after ACL reconstruction and may affect patient satisfaction and functional recovery. PRF is an autologous bioregenerative product with potential to support soft-tissue healing.

Objective: To determine whether PRF application at the donor site reduces anterior knee sensory deficit compared with standard surgical care.

Design and Participants: Single-center, prospective, pilot, non-randomized study with two parallel cohorts (PRF vs standard care). Competitively active male athletes meeting prespecified eligibility criteria are followed at 4, 8, and 12 months post-surgery. Recruitment window: January 2022 to January 2023.

Interventions: In the PRF cohort, PRF is prepared intraoperatively and applied to the donor site per manufacturer protocol; the comparator cohort receives standard closure without PRF.

Assessments:

Primary outcome: Proportion of participants without anterior knee sensory deficit at 12 months. Sensory testing is performed over a predefined 9-point area lateral to the surgical scar (eyes closed; contralateral knee used as reference if uncertain).

Secondary outcomes: Patient-reported knee function instruments (International Knee Documentation Committee [IKDC] Subjective Knee Form and Lysholm Knee Scoring Scale), each reported as total score (0-100; higher scores indicate better function) at 4, 8, and 12 months; optional MRI-based assessments of the donor site per protocol; safety monitoring of adverse events.

Analysis (planned): Group comparisons using appropriate categorical and non-parametric methods with prespecified approaches to handle multiplicity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Isolated anterior cruciate ligament rupture confirmed by MRI and clinical examination
* Planned ACL reconstruction with BPTB autograft
* Written informed consent provided

Exclusion Criteria:

* Previous knee surgery on the affected knee
* Associated ligament injuries requiring additional reconstruction
* Significant cartilage damage (Outerbridge grade III-IV beyond donor site changes)
* Systemic disease affecting wound healing (e.g., diabetes mellitus, autoimmune disease)
* Active infection
* Refusal or inability to provide informed consent

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing ACL reconstruction with bone-patellar tendon-bone (BPTB) autograft at the University Clinical Center of Serbia
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Proportion of participants without anterior knee sensory deficit at the donor site | 12 months post-surgery
  Sensory function assessed over a predefined 9-point area lateral to the surgical scar; deficit coded as 1 if >3 points are reported as "no or altered touch," otherwise 0. Assessment performed with eyes closed; contralateral knee used for reference if uncertain. Measure Type & Units: Percentage of participants (%)

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) Subjective Knee Form score (0-100; higher scores indicate better function) | Baseline, 4, 8, and 12 months post-surgery
  Patient-reported outcome; total score ranges from 0 (worst) to 100 (best).

OTHER OUTCOMES:
Lysholm Knee Scoring Scale (0-100; higher scores indicate better function) | Baseline, 4, 8, 12 months after surgery
  Patient-reported outcome; total score ranges from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center of Serbia (UKCS), Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy considerations and institutional regulations. Summary results will be published in peer-reviewed journals.

REFERENCES:
- [Background] Shichman I, Baruchi D, Rachevsky G, Amzallag N, Brandstetter AS, Vidra M, Morag G. Bone filling decreases donor site morbidity after anterior cruciate ligament reconstruction with bone-patellar tendon-bone autografts. Arch Orthop Trauma Surg. 2023 May;143(5):2565-2572. doi: 10.1007/s00402-022-04572-5. Epub 2022 Aug 2. PMID 35916963
- [Derived] Milovanovic D, Kadija M, Gavrilovic D, Sreckovic S, Bilanovic M, Matic A, Vukman P. Sensory Deficit Following Anterior Cruciate Ligament Reconstruction with Bone-Patellar Tendon-Bone Autograft: Platelet-Rich Fibrin (PRF) Could Provide a Solution. Medicina (Kaunas). 2025 Dec 12;61(12):2202. doi: 10.3390/medicina61122202. PMID 41470204
- Available data/document: Informed Consent Form: Ethics Committee approval No. — http://www.kcs.ac.rs/index.php/eticki-odbor

DOCUMENTS (3):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT07257666/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT07257666/SAP_001.pdf
  • Informed Consent Form (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT07257666/ICF_002.pdf